CLINICAL TRIAL: NCT06662331
Title: Effects of Low Medial Ramus Osteotomy Performed During Bilateral Sagittal Split Osteotomy on Neurosensorial Recovery During Post-Operative Period
Brief Title: Effects of Low Medial Ramus Osteotomy on Neurosensorial Recovery During Post-Operative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Törel Saygı (Other)
Responsible Party: Sponsor-Investigator, Ali Törel Saygı, Corresponding Author, Bezmialem Vakif University
Organization: Bezmialem Vakif University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 22/3
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Orthognathic Surgical Procedures
Keywords: orthognathic surgery; osteotomy modification

STUDY DESIGN:
Intervention Model Description: Double Blind
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hunsuck-Epker Modification (Experimental): A kind of ostoeotomy modification used during bilateral sagittal
  Interventions: Procedure: Bilateral Sagittal Split Osteotomy
- Low and short medial osteotomy (Experimental): A kind of ostoeotomy modification used during bilateral sagittal
  Interventions: Procedure: Bilateral Sagittal Split Osteotomy

INTERVENTIONS:
Procedure: Bilateral Sagittal Split Osteotomy — A surgical procedure to correct dentofacial deformities

SUMMARY:
The aim of this study is to compare the post-operative neurosensorial disturbances of Hunsuck-Epkerr and "low and short medial osteotomy" modifications of sagittal split ramus osteotomy. Patients at the ages of 18-35 with dentofacial deformity who applied for orthognathic surgery were included in the present study. The present study performed with split-mouth randomised controlled trial design, therefore osteotomies on one side were performed with Hunscuk-Epkerr modification and the contralateral side with low and short medial osteotomy modification. Double blinded evaluations of neuro sensorial alterations were performed at the 1st, 3rd and 6th months post-operatively. Painful stimuli, two-point discrimination, pressure and brush stroke direction tests were evaluated. Subjective neurosensorial recovery was also evaluated with VAS scores given by patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dentofacial deformity who needs orthognatic surgery

Exclusion Criteria:

* The patients with medical conditions that may affect the potential of nerve regeneration,
* The patient who need additional osteotomies such as genioplasty or mandibular subapical segmental osteotomies
* The patients with bad split or interrupted IAN
* The patients with more than 5 mm expected buccal osseous gap between proximal and distal segments

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Functional Sensory Recovery | 6 months
  Kind of scale, calculated with different neurosensorial investigation methods. Scored between S0-S4. S0 means total sensory loss, S4 means total sensory recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No